CLINICAL TRIAL: NCT01244347
Title: Randomized Clinical Trial to Evaluate the Efficacy of High Dose of Folic Acid to Prevent the Occurrence of Congenital Malformations
Brief Title: Folic Acid Dosage and Malformations Reduction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: International Centre of Birth Defects (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FARM 6KWTCT; 2008-004334-25 (EudraCT Number)
Record Dates: First submitted 2010-10-11; First posted 2010-11-19 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Congenital Malformations
Keywords: folic acid; malformations; prevention
MeSH Terms: conditions — Congenital Abnormalities | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- folic acid 4 mg (Experimental)
  Interventions: Drug: folic acid
- folic acid 0.4 mg (Active Comparator)
  Interventions: Drug: folic acid

INTERVENTIONS:
Drug: folic acid
  Arms: folic acid 4 mg
Drug: folic acid
  Arms: folic acid 0.4 mg

SUMMARY:
In 1991 the Medical Research Council Vitamin Study Group and in 1992 the Hungarian randomised clinical trial have shown conclusively that the risk of neural tube defects can be reduced substantially by taking folic acid during the peri-conceptional period. At present there is enough evidence to support the hypothesis that folic acid supplementation can reduce the risk of all congenital malformations or of a specific and selected group of them, namely: neural tube defects, oral clefts, cardiac defects, urinary tract anomalies except hypospadias, limb reduction defects, omphalocele, anal atresia and trisomy 21.

The hypothesis that a higher intake of folic acid is related to an higher risk reduction of neural tube defects and of other congenital malformations is the main rationale for the present study.

The present study is a randomized, double-blind, controlled trial evaluating whether supplementation with folic acid at high dose (4 mg/day) reduces the overall risk of major congenital malformations in the population more than the standard recommended dose (0.4 mg/day). At the enrolment visit all the eligible women will be interviewed to assess sociodemographic, life style and health status. After randomization, women will be interviewed every 4 months to evaluate pregnancy status. Women who have a pregnancy diagnosis during the study period will be interviewed by telephone at the expected 16, 24 and 40 weeks of gestation to evaluate the pregnancy outcome. The health status of live births will be evaluated at the child's age of 1 month, 3 months and 1 year.

The primary aim of this project is conducting a study to assess the effect of folic acid periconceptional supplementation of 4 mg/day compared to the 0.4 mg/day standard dose on reducing the occurrence of all congenital malformations. Secondary aims of this study include comparing severity of CMs in offspring of trial mothers, rates of "selected congenital malformations", rates of twinning, miscarriages, recurrent abortions, small-for-gestational age, preeclampsia and abruptio placentae. The sample size is not easy to be computed because lacking robust estimate of the size effect of the treatment. Three hypotheses of a size effect of 45%, 26% and 13% were considered. A sample size of outcomes (and women) respectively of 2,006 (5,015), 8,510 (21,275) and 30,126 (75,315) is needed. Since the sample size needed to evaluate different scenarios is large, the present study is also the pilot study to promote an international prospective meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 44 years
* women who intend to become pregnant (not excluded women

Exclusion Criteria:

* pregnant women
* women planning to move to an area where the study is not ongoing
* women who do not understand and speak Italian
* women who do not have a phone
* women affected by epilepsy, even not assuming anticonvulsivant drugs
* women affected by diabetes
* women who previously had a tumour or a disease relevant for the study (Crohn disease, rheumatoid arthritis, ulcerative colitis)
* women who recently assumed antifolates, like methotrexate
* women who currently abuse or previously abused alcohol
* obese women
* vegetarian women
* women who had a previous pregnancy with neural tube defect (NTD) or any other congenital structural defect
* women or partners with NTD, or one of their relatives with an NTD
* women with positive family history for breast or colorectal cancer
* women with positive family or personal history of hereditary syndrome like adenomatous polyposis, or hereditary nonpolyposis colorectal cancer
* women allergic to folic acid
* women presenting contraindications to folic acid
* women affected by megaloblastic anaemia
* assuming folic acid at defined doses for conditions other than those already mentioned

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5000 (Estimated)
Dates: Start 2009-07; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
number of congenital malformations | 112 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 28 weeks to all possible outcomes, plus 52 weeks of baby observation.

SECONDARY OUTCOMES:
rate of selected congenital malformations | 112 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 28 weeks to all possible outcomes, plus 52 weeks of baby observation.
Miscarriages and recurrent abortions | 47 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 15 weeks as a mean of time from conception to different clinical conditions related to miscarriage.
pre-eclampsia | 60 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 28 weeks to the occurrence of pre-eclampsia.
abruptio placentae | 34 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 34 weeks to the occurrence of abruptio placentae.
intrauterine growth restriction | 31 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 31 weeks to the occurrence of intrauterine growth restriction.
pre-term delivery | 30 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 30 weeks to the occurrence of pre-term delivery.
multiple births | 24 weeks
  The time frame was computed as an average of 32 weeks before conception, plus an average of 24 weeks to the possible diagnosis of twinnings or delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Bortolus, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona
Locations (32):
- Italy (32):
  - Ospedale di Adria, Adria, Rovigo
  - Ospedale San Luca, Trecenta, Rovigo
  - Ospedale di Conegliano, Conegliano, Treviso
  - Family Health Centre, Montebelluna, Treviso
  - Family Health Practice, Oderzo, Treviso
  - Family Health Practice, Villorba, Treviso
  - Ospedale Sant'Antonio Abate, Gallarate, Varese
  - Family Health Practice, Camponogara, Venezia
  - Family Health Centre, Martellago, Venezia
  - Family Health Practice, Mira, Venezia
  - Family Health Centre, Noale, Venezia
  - Family Health Centre, San Pietro di Stra, Venezia
  - Family Health Centre, Vogonovo, Venezia
  - Ospedale di Bussolengo, Bussolengo, Verona
  - Ospedale di Legnago, Legnago, Verona
  - Ospedale di San Bonifacio, San Bonifacio, Verona
  - Family Health Centre, Bassano, Vicenza
  - Ospedale San Bassiano, Bassano, Vicenza
  - General Practice, Dueville, Vicenza
  - General Practice, Malo, Vicenza
  - General Practice, Schio, Vicenza
  - General Practice, Sovizzo, Vicenza
  - Ospedale Boldrini, Thiene, Vicenza
  - Ospedale di Valdagno, Valdagno, Vicenza
  - Ospedale di Vicenza, Vicenza, VI
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Family Health Centre, Padua
  - Family Health Centre, Verona
  - General Practice, Verona
  - Ospedale Civile Maggiore, Verona
  - Policlinico G.B. Rossi, Verona

REFERENCES:
- [Background] Badovinac RL, Werler MM, Williams PL, Kelsey KT, Hayes C. Folic acid-containing supplement consumption during pregnancy and risk for oral clefts: a meta-analysis. Birth Defects Res A Clin Mol Teratol. 2007 Jan;79(1):8-15. doi: 10.1002/bdra.20315. PMID 17133404
- [Background] Berry RJ, Li Z, Erickson JD, Li S, Moore CA, Wang H, Mulinare J, Zhao P, Wong LY, Gindler J, Hong SX, Correa A. Prevention of neural-tube defects with folic acid in China. China-U.S. Collaborative Project for Neural Tube Defect Prevention. N Engl J Med. 1999 Nov 11;341(20):1485-90. doi: 10.1056/NEJM199911113412001. PMID 10559448
- [Background] Botto LD, Olney RS, Erickson JD. Vitamin supplements and the risk for congenital anomalies other than neural tube defects. Am J Med Genet C Semin Med Genet. 2004 Feb 15;125C(1):12-21. doi: 10.1002/ajmg.c.30004. PMID 14755429
- [Background] Catov JM, Bodnar LM, Ness RB, Markovic N, Roberts JM. Association of periconceptional multivitamin use and risk of preterm or small-for-gestational-age births. Am J Epidemiol. 2007 Aug 1;166(3):296-303. doi: 10.1093/aje/kwm071. Epub 2007 May 11. PMID 17496313
- [Background] Czeizel AE, Dudas I. Prevention of the first occurrence of neural-tube defects by periconceptional vitamin supplementation. N Engl J Med. 1992 Dec 24;327(26):1832-5. doi: 10.1056/NEJM199212243272602. PMID 1307234
- [Background] Ingrid Goh Y, Bollano E, Einarson TR, Koren G. Prenatal multivitamin supplementation and rates of congenital anomalies: a meta-analysis. J Obstet Gynaecol Can. 2006 Aug;28(8):680-689. doi: 10.1016/S1701-2163(16)32227-7. PMID 17022907
- [Background] Prevention of neural tube defects: results of the Medical Research Council Vitamin Study. MRC Vitamin Study Research Group. Lancet. 1991 Jul 20;338(8760):131-7. PMID 1677062
- [Derived] Bortolus R, Blom F, Filippini F, van Poppel MN, Leoncini E, de Smit DJ, Benetollo PP, Cornel MC, de Walle HE, Mastroiacovo P; Italian and Dutch folic acid trial study groups. Prevention of congenital malformations and other adverse pregnancy outcomes with 4.0 mg of folic acid: community-based randomized clinical trial in Italy and the Netherlands. BMC Pregnancy Childbirth. 2014 May 13;14:166. doi: 10.1186/1471-2393-14-166. PMID 24884885
- See also: Related Info — http://www.folictrial.org